CLINICAL TRIAL: NCT04079920
Title: BASELINE VARIABLES PREDICTING TREATMENT RESPONSE AT 6 MONTHS IN ADULT RHEUMATOID ARTHRITIS PATIENTS TREATED WITH TOFACITINIB 5MG BID IN A NON-INTERVENTIONAL SETTING (TREAT - RA)
Brief Title: Predictors of Response to Tofacitinib Treatment in Rheumatoid Arthritis Patients
Acronym: TREAT-RA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921342; TREAT-RA (Other: Alias Study Number)
Record Dates: First submitted 2019-08-05; First posted 2019-09-06 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
This is a 24-month, prospective, non-interventional, multi-center study with primary aim to identify baseline characteristics of patients that predict response at 6 months of treatment. The study also aims to describe the treatment patterns of RA patients prescribed tofacitinib in a real-world setting and assess the effect of treatment on patient quality of life and physical function. Finally the study will assess the use of healthcare resources and costs in patients with RA treated with tofacitinib in Greece.

The planned recruitment period is 12 months. The planned observation period of each patient is 12 months. In this time period up to 4 visits will be documented.

The study will be reviewed and approved by the Central Regulatory Committee for NIS and IRB Board of each participating site

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with moderately to severely active rheumatoid arthritis who start treatment with tofacitinib in usual clinical practice conditions in compliance with the label

  1. Patients aged ≥ 18 years
  2. Confirmed Diagnosis of Rheumatoid Arthritis by rheumatologist
  3. Patients with moderate to severe RA diagnosed according to local practice who have already been started on treatment with tofacitinib, for at most seven working days .
  4. Patients eligible for tofacitinib treatment according to current approved Summary of Product Characteristics (SmPC).
  5. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients meeting any of the following criteria will not be included in the study:

  1. Exclusion Criteria according to the Xeljanz® SmPC.
  2. Contraindications to Xeljanz® according to SmPC.
  3. Hypersensitivity to the active substance (tofacitinib) or to any of the excipients.
  4. Active tuberculosis (TB), serious infections, such as sepsis, or opportunistic infections.
  5. Receipt of any investigational drug within 3 months before study inclusion as well as currently not participating in an interventional clinical trial.
  6. Subjects who have received any previous treatment with tofacitinib or other JAK inhibitors.
  7. Subjects who are investigational site staff members or subjects who are Pfizer employees directly involved in the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting in outpatient clinics of Hospitals in Greece (secondary care)
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Greece (17):
  - University General Hospital of Athens "Attikon", Athens, Attica
  - 251 Air Force Hospital of Athens, Athens
  - General Hospital of Athens Gennimatas, Athens
  - Ippokrateio General Hospital of Athens, Athens
  - Laiko General Hospital of Athens, Athens
  - Naval Hospital of Athens, Athens
  - Nearchou 18, Crete
  - Univerisity General Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - KAT General Hospital of Attica, Kfisia
  - Univerisity General Hospital of Larisa, Larissa
  - University General Hospital of Patras, Pátrai
  - Agios Andreas General Hospital of Patra, Pátrai
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - Euromedica Kyanous Stavros General Clinic, Thessaloniki
  - General Hospital of Thessaloniki Ippokrateio, Thessaloniki
  - Asklipieio General Hospital of Voula, Voula

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with moderate-to-severe active rheumatoid arthritis who initiated tofacitinib in real-world and in a non-interventional setting in Greece were observed in this study.
Groups:
- Tofacitinib: Participants with rheumatoid arthritis who were treated with tofacitinib in usual clinical practice conditions (outpatient clinics of hospitals) in compliance with the current approved summary of product characteristics (SmPC) were observed in this study. The recommended dosage was tofacitinib 5 milligrams (mg) tablet twice daily.
Period: Overall Study
Arm/Group | Tofacitinib
Started | 198
Completed | 150
Not Completed | 48
Not completed — Adverse event, not related to study drug | 2
Not completed — Adverse event related to study drug | 10
Not completed — Death | 2
Not completed — Lost to Follow-up | 22
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 11

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements.
Groups:
- Tofacitinib: Participants with rheumatoid arthritis who were treated with tofacitinib in usual clinical practice conditions (outpatient clinics of hospitals) in compliance with the current approved SmPC were observed in this study. The recommended dosage was tofacitinib 5 mg tablet twice daily.
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (11.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission and Low Disease Activity (LDA) at Month 6 Assessed Using 28-Joint Disease Activity Score C-Reactive Protein (DAS28-4 CRP)
Description: Remission is defined as DAS28-4 CRP less than (<) 2.6 and DAS28-4 CRP < 3.2 corresponds to LDA. DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). It includes components: tender joint count (TJC) and swollen joint count ((SJC) [both out of 28 evaluated joints], CRP milligram per liter (mg/l) and Patient's Global Assessment of Arthritis Disease Activity (PtGA) recorded on 100 millimeter (mm) visual analogue scale (VAS) (scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). DAS28-4 CRP is calculated as: 0.56 * square root (sqrt) (TJC) + 0.28 * sqrt (SJC) + 0.36 * ln (CRP+1) + 0.014*PtGA + 0.96; where ln = natural logarithm.
Time Frame: Month 6
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. Here, "Number of Participants Analyzed" signifies number of participants evaluable and who contributed to data for this outcome measure. Missing components were imputed by carrying forward the last non-missing post-baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 152
Percentage of participants
  Remission | 29.6
  LDA | 41.4

2. Secondary Outcome: Percentage of Participants With Remission and LDA at Month 12 Assessed Using DAS28-4 CRP
Description: Remission is defined as DAS28-4 CRP < 2.6 and DAS28-4 CRP < 3.2 corresponds to LDA. DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). It includes components: TJC and SJC assessed using 28 joints, CRP (mg/l) and PtGA recorded on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). DAS28-4 CRP is calculated as: 0.56 * (sqrt) (TJC28) + 0.28 * sqrt (SJC28) + 0.36 * ln (CRP+1) + 0.014*PtGA + 0.96; where ln = natural logarithm.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 150
Percentage of participants
  Remission | 33.3
  LDA | 55.3

3. Secondary Outcome: Change From Baseline in DAS28-4 (ESR) and DAS28-4 (CRP)
Description: DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). It includes components: TJC and SJC both assessed using 28 joints, CRP (mg/l) and PtGA recorded recorded on VAS scores (mm). DAS28-4 CRP is calculated as: 0.56 * sqrt (TJC28) + 0.28 * sqrt (SJC28) + 0.36 * ln (CRP+1) + 0.014*PtGA + 0.96; where ln = natural logarithm. DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). It includes components: TJC and SJC both assessed using 28 joints, ESR using mm/ hour and PtGA in recorded on VAS (mm). DAS28-4 ESR is calculated as: 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.70*In (ESR) + 0.014*PtGA where In = natural logarithm. The calculated range of DAS28-4 CRP and DAS 28-4 ESR is 0 (no disease activity) to 10 (maximal disease activity). A decrease from baseline in score indicates improvement of disease activity.
Time Frame: Baseline, Months 3, 6 and 12
Population: FAS population was analyzed. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. "Number Analyzed" signifies number of participants evaluable at specified time points. Missing components were imputed by carrying forward the last non-missing post-baseline value.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 192
Units on a scale
  Change at Month 3: DAS28-4(CRP): number analyzed (Participants) | 158
  Change at Month 3: DAS28-4(CRP) | -1.25 (1.38)
  Change at Month 6: DAS28-4(CRP): number analyzed (Participants) | 145
  Change at Month 6: DAS28-4(CRP) | -1.47 (1.40)
  Change at Month 12: DAS28-4(CRP): number analyzed (Participants) | 144
  Change at Month 12: DAS28-4(CRP) | -1.73 (1.46)
  Change at Month 3: DAS 28-4 (ESR): number analyzed (Participants) | 169
  Change at Month 3: DAS 28-4 (ESR) | -1.15 (1.47)
  Change at Month 6:DAS 28-4 (ESR): number analyzed (Participants) | 147
  Change at Month 6:DAS 28-4 (ESR) | -1.42 (1.58)
  Change at Month 12: DAS 28-4 (ESR): number analyzed (Participants) | 146
  Change at Month 12: DAS 28-4 (ESR) | -1.58 (1.61)

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Months 3, 6 and 12
Description: HAQ-DI is a participant-reported assessment which assess the degree of difficulty a participant had experienced during the last week in 8 domains/categories of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 items. Each item is scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Any activity requiring assistance from another individual or the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranges from 0 to 3, where 0 indicates least difficulty and 3 indicates extreme difficulty.
Time Frame: Baseline, Months 3, 6 and 12
Population: FAS population was analyzed. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to table; however, may not have evaluable data for every row. "Number Analyzed" signifies number of participants evaluable at specified time points. If one or two domains had missing data, score was calculated as: sum of non-missing domain scores/number of non-missing domains.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 190
Units on a scale
  Change at Month 3: number analyzed (Participants) | 159
  Change at Month 3 | -0.25 (0.56)
  Change at Month 6: number analyzed (Participants) | 138
  Change at Month 6 | -0.40 (0.60)
  Change at Month 12: number analyzed (Participants) | 122
  Change at Month 12 | -0.40 (0.60)

5. Secondary Outcome: Number of Participants With Remission According to Simplified Disease Activity Index (SDAI) <=3.3 at Months 3, 6, and 12
Description: Remission is defined as SDAI <=3.3. SDAI is a composite end point, calculated at each time point using the formula: as TJC + SJC both assessed using 28 joints + PtGA (assessed on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity) + Physician's Global Assessment of Health [PhGA] (assessed on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity)+ CRP (mg/dL).
Time Frame: Months 3, 6 and 12
Population: FAS population was analyzed. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with SDAI at specified time points. No imputation was applied for missing values in any visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 190
Participants
  Month 3: number analyzed (Participants) | 164
  Month 3 | 12
  Month 6: number analyzed (Participants) | 142
  Month 6 | 14
  Month 12: number analyzed (Participants) | 140
  Month 12 | 22

6. Secondary Outcome: Number of Participants With Remission According to Clinical Disease Activity Index (CDAI) <=2.8 at Months 3, 6, and 12
Description: Remission is defined as CDAI <=2.8. CDAI is a composite end point, calculated based on each time-point using TJC + SJC both assessed using 28 joints + PtGA (assessed on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity) + PhGA (assessed on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity).
Time Frame: Months 3, 6 and 12
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with CDAI at specified time points. No imputation was applied for missing values in any visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Participants
  Month 3: number analyzed (Participants) | 172
  Month 3 | 11
  Month 6: number analyzed (Participants) | 152
  Month 6 | 16
  Month 12: number analyzed (Participants) | 150
  Month 12 | 24

7. Secondary Outcome: Number of Participants With Remission According to DAS28-4 ESR<2.6 at Months 3, 6, and 12
Description: DAS28-4 ESR is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). Components includes: TJC, SJC both assessed using 28 joints, ESR (mm/h) and PtGA (mm) (recorded on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher score indicates high disease activity). The calculation of DAS28-4 ESR is as follows: 0.56 * sqrt (TJC28) + 0.28 * sqrt (SJC28) + 0.70* In (ESR) + 0.014* (PtGA); where ln = natural logarithm. DAS28-4 (ESR) score of <2.6 indicates remission.
Time Frame: Months 3, 6 and 12
Population: FAS population was analyzed. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with DAS 28-4 (ESR) at specified time points. No imputation was applied for missing values in any visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 192
Participants
  Month 3: number analyzed (Participants) | 165
  Month 3 | 25
  Month 6: number analyzed (Participants) | 144
  Month 6 | 30
  Month 12: number analyzed (Participants) | 141
  Month 12 | 40

8. Secondary Outcome: Number of Participants With Remission According to DAS28-4 CRP <2.6 at Months 3, 6, and 12
Description: DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). Components includes: TJC, SJC both assessed using 28 joints, CRP (mg/l) and PtGA (mm) (recorded on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher score indicates high disease activity). The calculation of DAS28-4 CRP is as follows: 0.56 * sqrt (TJC) + 0.28 * sqrt (SJC) + 0.36 * ln (CRP+1) + 0.014*PtGA + 0.96; where ln = natural logarithm. DAS28-4 (CRP) score of <2.6 indicates remission.
Time Frame: Months 3, 6 and 12
Population: FAS population was analyzed. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with DAS28-4 (CRP) at specified time points. No imputation was applied for missing values in any visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 190
Participants
  Month 3: number analyzed (Participants) | 164
  Month 3 | 31
  Month 6: number analyzed (Participants) | 142
  Month 6 | 45
  Month 12: number analyzed (Participants) | 140
  Month 12 | 49

9. Secondary Outcome: Number of Participants With LDA According to SDAI <=11 at Months 3, 6, and 12
Description: LDA is defined as SDAI <=11. SDAI is a composite end point, calculated at each time point using the formula: as TJC + SJC (both assessed using 28 joints) + PtGA (assessed on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity) + PhGA (assessed on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity)+ CRP (mg/dL).
Time Frame: Months 3, 6 and 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 190
Participants
  Month 3: number analyzed (Participants) | 164
  Month 3 | 54
  Month 6: number analyzed (Participants) | 142
  Month 6 | 63
  Month 12: number analyzed (Participants) | 140
  Month 12 | 74

10. Secondary Outcome: Number of Participants With LDA According to CDAI <=10 at Months 3, 6, and 12
Description: LDA is defined as CDAI <=10. CDAI is a composite end point, calculated based on each time-point using TJC + SJC (both assessed using 28 joints) + PtGA (assessed on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity) + PhGA (assessed on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity.
Time Frame: Months 3, 6 and 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Participants
  Month 3: number analyzed (Participants) | 172
  Month 3 | 56
  Month 6: number analyzed (Participants) | 152
  Month 6 | 61
  Month 12: number analyzed (Participants) | 150
  Month 12 | 73

11. Secondary Outcome: Number of Participants With LDA According to DAS28-4 ESR (<3.2) at Months 3, 6, and 12
Description: DAS28-4 ESR is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). Components includes: TJC, SJC (both assessed using 28 joints), ESR (mm/h) and PtGA (recorded on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher score indicates high disease activity). The calculation of DAS28-4 ESR is as follows: 0.56 * sqrt (TJC28) + 0.28 * sqrt (SJC28) + 0.70* In(ESR) + 0.014* (PtGA); where ln = natural logarithm. DAS28-4 (ESR) score of <3.2 indicates LDA.
Time Frame: Months 3, 6 and 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 192
Participants
  Month 3: number analyzed (Participants) | 165
  Month 3 | 46
  Month 6: number analyzed (Participants) | 144
  Month 6 | 62
  Month 12: number analyzed (Participants) | 141
  Month 12 | 65

12. Secondary Outcome: Number of Participants With LDA According to DAS28-4 CRP<=3.2 at Months 3, 6, and 12
Description: LDA is defined as DAS28-4(CRP) score of <3.2. DAS28-4 CRP is a composite endpoint, calculated using 4 variables (represented by '-4' in the name). It includes components: TJC, SJC (both assessed using 28 joints), CRP (mg/l) and PtGA (mm) (recorded on 100 mm VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity). The calculation of DAS28-4 CRP is as follows: 0.56*sqrt (TJC) + 0.28*sqrt (SJC) + 0.36*ln (CRP+1) + 0.014*PtGA + 0.96; where ln = natural logarithm. DAS28-4 (CRP) score of <3.2 indicates LDA.
Time Frame: Months 3, 6 and 12
Population: FAS population was analyzed. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with DAS 28-4 (CRP) at specified time points. No imputation was applied for missing values in any visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 190
Participants
  Month 3: number analyzed (Participants) | 164
  Month 3 | 59
  Month 6: number analyzed (Participants) | 142
  Month 6 | 63
  Month 12: number analyzed (Participants) | 140
  Month 12 | 82

13. Secondary Outcome: Percentage of Participants Achieving HAQ-DI Response at Months 3,6 and 12
Description: HAQ-DI is a participant-reported assessment which assess the degree of difficulty a participant had experienced during the last week in 8 domains/categories of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2 to 3 items. Each item is scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Any activity requiring assistance from another individual or the use of an assistive device adjusts to a minimum score of 2 to represent a more limited functional status. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranges from 0 to 3, where 0 indicates least difficulty and 3 indicates extreme difficulty. A HAQ-DI response is defined as a decrease from baseline of at least 0.22.
Time Frame: Months 3, 6 and 12
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 190
Percentage of participants
  Month 3: number analyzed (Participants) | 159
  Month 3 | 56.6
  Month 6: number analyzed (Participants) | 138
  Month 6 | 65.9
  Month 12: number analyzed (Participants) | 122
  Month 12 | 71.3

14. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQol) -5 Dimensions (EQ-5D) Health State Profile at Months 3, 6 and 12
Description: EQ-5D is a standardized instrument used to measure quality of life. It is based on five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three responses and the participant is asked to select the response that best describes them. The responses are scored 1-3 where 1 indicates no problems, 2 indicates some problems and 3 indicates unable to perform normal activities. The score (1 to 3), for each dimension is weighted based on United Kingdom (UK) data (Dolan et al 1995). An algorithm was applied to calculate the total EQ-5D health state score. Maximum and minimum score value were 1 and -0.6 respectively. Higher score indicates better health state.
Time Frame: Baseline, Months 3, 6 and 12
Population: FAS population was analyzed. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with EQ-5D score at specified time points. Missing weighted dimension scores were replaced by the mean of non-missing ones.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 193
Units on a scale
  Change at Month 3: number analyzed (Participants) | 171
  Change at Month 3 | 0.18 (0.02)
  Change at Month 6: number analyzed (Participants) | 145
  Change at Month 6 | 0.23 (0.02)
  Change at Month 12: number analyzed (Participants) | 141
  Change at Month 12 | 0.23 (0.02)

15. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Questionnaire Score at Months 3, 6 and 12
Description: FACIT-fatigue questionnaire score consists of 13 self-evaluated questions. Each question is scored from 0 to 4; the sum of all responses resulted in the FACIT-fatigue score of 0 (maximum fatigue) to 52 (no fatigue). A higher score represents better participant status.
Time Frame: Baseline, Months 3, 6 and 12
Population: FAS population was analyzed. All participants reported under "Number of Participants analyzed" =number of participant evaluable and contributed data to table; however, may not have evaluable data for every row. "Number Analyzed"=number of participants evaluable at specified time points. If more than 50% of the items were non-missing, then score was prorated by multiplying the sum of the subscale by the number of items in the subscale, then dividing by the number of items actually answered.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib
Number analyzed (Participants) | 195
Units on a scale
  Change at Month 3: number analyzed (Participants) | 172
  Change at Month 3 | 6.8 (0.66)
  Change at Month 6: number analyzed (Participants) | 145
  Change at Month 6 | 7.21 (0.65)
  Change at Month 12: number analyzed (Participants) | 144
  Change at Month 12 | 8.71 (0.66)

16. Secondary Outcome: Change From Baseline in Mean Duration of Morning Stiffness at Day 1 and 2 of Months 3, 6 and 12
Description: The duration of morning stiffness is determined by asking the following questions: "Over the last 2 days, when did you wake in the morning? Over the last 2 days, when were you able to resume your normal activities without stiffness?". Time elapsed when participant woke up in morning and was able to resume normal activities without stiffness in minutes.
Time Frame: Baseline, Day 1 and 2 of Months 3, 6 and 12
Population: FAS population was analyzed. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants with morning stiffness evaluable at specified time points. No imputation was applied for missing values in any visit.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tofacitinib
Number analyzed (Participants) | 153
Minutes
  Change at Month 3: Day 1: number analyzed (Participants) | 128
  Change at Month 3: Day 1 | -25.7 (43.02)
  Change at Month 6: Day 1: number analyzed (Participants) | 113
  Change at Month 6: Day 1 | -29.9 (42.68)
  Change at Month 12: Day 1: number analyzed (Participants) | 110
  Change at Month 12: Day 1 | -34.2 (44.27)
  Change at Month 3: Day 2: number analyzed (Participants) | 117
  Change at Month 3: Day 2 | -30.42 (46.9)
  Change at Month 6: Day 2: number analyzed (Participants) | 103
  Change at Month 6: Day 2 | -33.8 (43.50)
  Change at Month 12: Day 2: number analyzed (Participants) | 101
  Change at Month 12: Day 2 | -37.04 (41.89)

17. Secondary Outcome: Change From Baseline in the Work Productivity and Activity Impairment (WPAI) Questionnaire at Months 3, 6 and 12
Description: WPAI: 6-item questionnaire & scores are derived for four domains:absenteeism, presenteeism,work productivity loss & activity impairment.Question (Q)2 asked participants to indicate number of hours missed due to health problems in past 7 days. Q4 asked participants to indicate number of hours they worked in past 7 days.Q5 asked participants the degree to which their health affected productivity while working in past 7 days,on scale ranging from 0-10, Where 0 = health problems had no effect on their work & 10=health problems completely prevented participant from working. Q6 asked participants to indicate the degree to which their health affected their regular activities in past 7 days.Absenteeism=(Q2/[Q2 + Q4])*100.Presenteeism=(Q5/10)*100.Work Production Loss={(Q2/[Q2 + Q4])+(1-[Q2/(Q2 + Q4))*(Q5/10 )]}*100.Activity Impairment=(Q6/10)*100.Each WPAI domain is expressed as impairment percentages ranging from 0 to 100,with higher numbers indicating greater impairment &less productivity.
Time Frame: Baseline, Months 3, 6 and 12
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. All participants reported under "Number of Participants Analyzed" contributed data to table; however, may not have evaluable data for every row. Here, "Number Analyzed"= number of participants evaluable at specified time points.
Measure: Least Squares Mean (Standard Error); unit: Percentage of impairment
Arm/Group | Tofacitinib
Number analyzed (Participants) | 184
Percentage of impairment
  Change in Absenteeism: Month 3: number analyzed (Participants) | 54
  Change in Absenteeism: Month 3 | 3.9 (1.4)
  Change in Absenteeism: Month 6: number analyzed (Participants) | 47
  Change in Absenteeism: Month 6 | 1.7 (1.6)
  Change in Absenteeism: Month 12: number analyzed (Participants) | 50
  Change in Absenteeism: Month 12 | -0.08 (1.5)
  Change in Presenteeism: Month 3: number analyzed (Participants) | 67
  Change in Presenteeism: Month 3 | 4.0 (2.8)
  Change in Presenteeism: Month 6: number analyzed (Participants) | 65
  Change in Presenteeism: Month 6 | 4.2 (3.6)
  Change in Presenteeism: Month 12: number analyzed (Participants) | 55
  Change in Presenteeism: Month 12 | 2.8 (3.8)
  Change in Work Production Loss: Month 3: number analyzed (Participants) | 53
  Change in Work Production Loss: Month 3 | 0.2 (3.1)
  Change in Work Production Loss: Month 6: number analyzed (Participants) | 47
  Change in Work Production Loss: Month 6 | -1.9 (3.7)
  Change in Work Production Loss: Month 12: number analyzed (Participants) | 48
  Change in Work Production Loss: Month 12 | -1.9 (3.6)
  Change in Activity Impairment: Month 3: number analyzed (Participants) | 161
  Change in Activity Impairment: Month 3 | 5.1 (1.8)
  Change in Activity Impairment: Month 6: number analyzed (Participants) | 141
  Change in Activity Impairment: Month 6 | 7.6 (2.2)
  Change in Activity Impairment: Month 12: number analyzed (Participants) | 140
  Change in Activity Impairment: Month 12 | 10.3 (2.3)

18. Secondary Outcome: Percentage of Participants With Treatment Satisfaction at Baseline and Month 12
Description: Participant's satisfaction with treatment was assessed on a 5-point scale (where 0 = very dissatisfied and 4 = very satisfied) in response to the question "How satisfied are you with the drugs you received for your arthritis during the last year?"
Time Frame: Baseline, Month 12
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. No imputation was applied for missing values in any visit. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Percentage of participants
  Baseline: Very dissatisfied | 13.6
  Baseline: Somewhat dissatisfied | 34.3
  Baseline: Neither satisfied nor dissatisfied | 31.8
  Baseline: Somewhat satisfied | 17.7
  Baseline: Very satisfied | 2.5
  Month 12: Very dissatisfied: number analyzed (Participants) | 150
  Month 12: Very dissatisfied | 2.0
  Month 12: Somewhat dissatisfied: number analyzed (Participants) | 150
  Month 12: Somewhat dissatisfied | 4.7
  Month 12: Neither satisfied nor dissatisfied: number analyzed (Participants) | 150
  Month 12: Neither satisfied nor dissatisfied | 16.7
  Month 12: Somewhat satisfied: number analyzed (Participants) | 150
  Month 12: Somewhat satisfied | 46.0
  Month 12: Very satisfied: number analyzed (Participants) | 150
  Month 12: Very satisfied | 30.7

19. Secondary Outcome: Patient Global Assessment (PtGA) at Baseline, Months 3, 6 and 12
Description: PtGA of Arthritis was measured using a VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity in response to the question "Considering all the way your arthritis affects you, how are you feeling today?".
Time Frame: Baseline, Months 3, 6 and 12
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. Here, "Number Analyzed" signifies number of participants evaluable with PtGA score at specified time points. No imputation was applied for missing values in any visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
mm
  Baseline | 59.0 (23.43)
  Month 3: number analyzed (Participants) | 172
  Month 3 | 39.2 (23.60)
  Month 6: number analyzed (Participants) | 152
  Month 6 | 35.8 (23.65)
  Month 12: number analyzed (Participants) | 150
  Month 12 | 31.0 (21.56)

20. Secondary Outcome: Physician Global Assessment (PhGA) at Baseline, Months 3, 6 and 12
Description: PhGA was measured using a VAS scores ranging 0 [no disease activity] to 100 mm [maximum disease activity], higher scores=more disease activity in response to how the physician assesses the participant's overall arthritis at the time of the visit. This is an evaluation based on the participant's disease signs, functional capacity and physical examination, and should be independent of the PtGA of arthritis.
Time Frame: Baseline, Months 3, 6 and 12
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. Here, "Number Analyzed" signifies number of participants evaluable with PhGA score at specified time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
mm
  Baseline | 59.6 (19.8)
  Month 3: number analyzed (Participants) | 172
  Month 3 | 35.9 (21.93)
  Month 6: number analyzed (Participants) | 152
  Month 6 | 30.0 (20.73)
  Month 12: number analyzed (Participants) | 150
  Month 12 | 27.1 (21.26)

21. Secondary Outcome: Number of Participants as Per Treatment Received
Description: Number of participants who received tofacitinib as monotherapy,tofacitinib in combination therapy, tofacitinib switched from monotherapy to combination therapy, tofacitinib switched from combination therapy to monotherapy, tofacitinib in combination with disease modifying antirheumatic drugs (DMARD) then switched to tofacitinib monotherapy and tofacitinib in combination with DMARD then discontinued are presented in this outcome measure.
Time Frame: Up to 12 months
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Participants
  Tofacitinib as Monotherapy | 59
  Tofacitinib in Combination Therapy | 113
  Tofacitinib Switched From Monotherapy to Combination Therapy | 1
  Tofacitinib Switched From Combination Therapy to Monotherapy | 5
  Tofacitinib in Combination with DMARD Then Switched to Tofacitinib Monotherapy | 2
  Tofacitinib in Combination with DMARD Then Discontinued | 18

22. Secondary Outcome: Median Number of Visits to Rheumatologist or Other Rheumatoid Arthritis (RA) Specialist Since Last Visit
Description: The study consisted of 4 visits. Baseline (visit 1), Month 3 (visit 2), Month 6 (visit 3), Month 12 (final or close out visit). The number of visits to a rheumatologist or other RA specialist since the last visit were reported in this outcome measure.
Time Frame: Months 3, 6 and 12
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Median (Full Range); unit: Visits
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Visits
  Month 3: number analyzed (Participants) | 152
  Month 3 | 0.0 [0 to 5]
  Month 6: number analyzed (Participants) | 125
  Month 6 | 0.0 [0 to 3]
  Month 12: number analyzed (Participants) | 113
  Month 12 | 1.0 [0 to 5]

23. Secondary Outcome: Number of Participants With Diagnostic Test Since Last Visit
Description: The study consisted of 4 visits. Baseline (visit 1), Month 3 (visit 2), Month 6 (visit 3), Month 12 (final or close out visit). Number of participants who underwent the diagnostic tests since last visit including: whole blood cell (WBC), ESR/CRP, glucose, hepatic enzymes, urea, creatinine, lipid profile (total cholesterol [TC], low density lipoprotein [LDL], high density lipoprotein [HDL], triglycerides [TG]), X-rays, others are presented.
Time Frame: Months 3, 6 and 12
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Participants
  Month 3: number analyzed (Participants) | 174
  Month 3 | 76
  Month 6: number analyzed (Participants) | 152
  Month 6 | 59
  Month 12: number analyzed (Participants) | 150
  Month 12 | 50

24. Secondary Outcome: Number of Participants According to the Type of Diagnostic Test
Description: The study consisted of 4 visits. Baseline (visit 1), Month 3 (visit 2), Month 6 (visit 3), Month 12 (final or close out visit). Number of participants who underwent the diagnostic tests including: WBC, ESR/CRP, glucose, hepatic enzymes, urea, creatinine, lipid profile (TC,LDL,HDL,TG), X-rays, others summarized by visit are presented.
Time Frame: Months 3, 6 and 12
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Participants
  WBC- Month 3: number analyzed (Participants) | 76
  WBC- Month 3 | 69
  WBC- Month 6: number analyzed (Participants) | 59
  WBC- Month 6 | 50
  WBC- Month 12: number analyzed (Participants) | 50
  WBC- Month 12 | 42
  ESR- Month 3: number analyzed (Participants) | 76
  ESR- Month 3 | 69
  ESR- Month 6: number analyzed (Participants) | 59
  ESR- Month 6 | 55
  ESR- Month 12: number analyzed (Participants) | 50
  ESR- Month 12 | 48
  CRP- Month 3: number analyzed (Participants) | 76
  CRP- Month 3 | 67
  CRP- Month 6: number analyzed (Participants) | 59
  CRP- Month 6 | 55
  CRP- Month 12: number analyzed (Participants) | 50
  CRP- Month 12 | 47
  Glucose- Month 3: number analyzed (Participants) | 76
  Glucose- Month 3 | 56
  Glucose- Month 6: number analyzed (Participants) | 59
  Glucose- Month 6 | 44
  Glucose- Month 12: number analyzed (Participants) | 50
  Glucose- Month 12 | 39
  Hepatic enzymes- Month 3: number analyzed (Participants) | 76
  Hepatic enzymes- Month 3 | 66
  Hepatic enzymes- Month 6: number analyzed (Participants) | 59
  Hepatic enzymes- Month 6 | 49
  Hepatic enzymes- Month 12: number analyzed (Participants) | 50
  Hepatic enzymes- Month 12 | 44
  Urea- Month 3: number analyzed (Participants) | 76
  Urea- Month 3 | 62
  Urea- Month 6: number analyzed (Participants) | 59
  Urea- Month 6 | 48
  Urea- Month 12: number analyzed (Participants) | 50
  Urea- Month 12 | 44
  Creatinine- Month 3: number analyzed (Participants) | 76
  Creatinine- Month 3 | 63
  Creatinine- Month 6: number analyzed (Participants) | 59
  Creatinine- Month 6 | 50
  Creatinine- Month 12: number analyzed (Participants) | 50
  Creatinine- Month 12 | 44
  Lipid profile (TC, LDL, HDL, TG)- Month 3: number analyzed (Participants) | 76
  Lipid profile (TC, LDL, HDL, TG)- Month 3 | 29
  Lipid profile (TC, LDL, HDL, TG)- Month 6: number analyzed (Participants) | 59
  Lipid profile (TC, LDL, HDL, TG)- Month 6 | 37
  Lipid profile (TC, LDL, HDL, TG)- Month 12: number analyzed (Participants) | 50
  Lipid profile (TC, LDL, HDL, TG)- Month 12 | 29
  X-rays- Month 3: number analyzed (Participants) | 76
  X-rays- Month 3 | 1
  X-rays- Month 6: number analyzed (Participants) | 59
  X-rays- Month 6 | 4
  X-rays- Month 12: number analyzed (Participants) | 50
  X-rays- Month 12 | 3
  Others- Month 3: number analyzed (Participants) | 76
  Others- Month 3 | 13
  Others- Month 6: number analyzed (Participants) | 59
  Others- Month 6 | 8
  Others- Month 12: number analyzed (Participants) | 50
  Others- Month 12 | 4

25. Secondary Outcome: Number of Diagnostic Tests Since Last Visit
Description: The study consisted of 4 visits. Baseline (visit 1), Month 3 (visit 2), Month 6 (visit 3), Month 12 (final or close out visit). Diagnostic tests performed were as follow: WBC, ESR/CRP, glucose, hepatic enzymes, urea, creatinine, lipid profile (TC, LDL, HDL, TG), X-rays, others summarized by visit are presented.
Time Frame: Months 3, 6 and 12
Population: as for outcome 22
Measure: Number; unit: Diagnostic tests
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Diagnostic tests
  Month 3: number analyzed (Participants) | 174
  Month 3 | 488
  Month 6: number analyzed (Participants) | 152
  Month 6 | 292
  Month 12: number analyzed (Participants) | 150
  Month 12 | 323

26. Secondary Outcome: Number of Participants Hospitalized Since Last Visit
Description: The study consisted of 4 visits. Baseline (visit 1), Month 3 (visit 2), Month 6 (visit 3), Month 12 (final or close out visit). Number of participants hospitalized since their last visit were reported in this outcome measure.
Time Frame: Months 3, 6 and 12
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 198
Participants
  Month 3: number analyzed (Participants) | 174
  Month 3 | 3
  Month 6: number analyzed (Participants) | 152
  Month 6 | 0
  Month 12: number analyzed (Participants) | 150
  Month 12 | 1

27. Secondary Outcome: Number of Participants Hospitalized in Daycare and Night Care Since Last Visit
Description: The study consisted of 4 visits. Baseline (visit 1), Month 3 (visit 2), Month 6 (visit 3), Month 12 (final or close out visit). Number of participants hospitalized in daycare and nightcare since their last visit were reported in this outcome measure.
Time Frame: Months 3, 6 and 12
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 3
Participants
  Participants Hospitalized With Daycare: Month 3 | 0
  Participants Hospitalized With Daycare: Month 6: number analyzed (Participants) | 0
  Participants Hospitalized With Daycare: Month 12: number analyzed (Participants) | 1
  Participants Hospitalized With Daycare: Month 12 | 0
  Participants Hospitalized With Overnight Stay: Month 3 | 3
  Participants Hospitalized With Overnight Stay: Month 6: number analyzed (Participants) | 0
  Participants Hospitalized With Overnight Stay: Month 12: number analyzed (Participants) | 1
  Participants Hospitalized With Overnight Stay: Month 12 | 1

28. Secondary Outcome: Mean Number of Days Participants Were Hospitalized Since Last Visit
Description: The study consisted of 4 visits. Baseline (visit 1), Month 3 (visit 2), Month 6 (visit 3), Month 12 (final or close out visit). Mean number of days participants were hospitalized since last visit were reported in this outcome measure.
Time Frame: Baseline, Months 3, 6 and 12
Population: FAS population included participants who met the eligibility criteria, received at least one dose of tofacitinib and had at least one set of post-baseline measurements. "Number of Participants analyzed" signifies number of participant evaluable for this outcome measure. "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tofacitinib
Number analyzed (Participants) | 3
Days
  Month 3 | 6.7 (2.1)
  Month 6: number analyzed (Participants) | 0
  Month 12: number analyzed (Participants) | 0

29. Secondary Outcome: Number of Participants According to Reason for Hospitalization Since Last Visit
Description: The study consisted of 4 visits. Baseline (visit 1), Month 3 (visit 2), Month 6 (visit 3), Month 12 (final or close out visit). Number of participants according to reason for hospitalization: polyarthritis, RA and pericarditis, RA flare, and right knee arthroplasty due to osteoarthritis since their last visit is presented in this outcome measure.
Time Frame: Months 3, 6 and 12
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib
Number analyzed (Participants) | 3
Participants
  Polyarthritis: Month 3 | 1
  Polyarthritis: Month 6: number analyzed (Participants) | 0
  Polyarthritis: Month 12: number analyzed (Participants) | 1
  Polyarthritis: Month 12 | 0
  RA and Pericarditis: Month 3 | 1
  RA and Pericarditis: Month 6: number analyzed (Participants) | 0
  RA and Pericarditis: Month 12: number analyzed (Participants) | 1
  RA and Pericarditis: Month 12 | 0
  RA flare: Month 3 | 1
  RA flare: Month 6: number analyzed (Participants) | 0
  RA flare: Month 12: number analyzed (Participants) | 1
  RA flare: Month 12 | 0
  Right knee arthroplasty due to Osteoarthritis: Month 3 | 0
  Right knee arthroplasty due to Osteoarthritis: Month 6: number analyzed (Participants) | 0
  Right knee arthroplasty due to Osteoarthritis: Month 12: number analyzed (Participants) | 1
  Right knee arthroplasty due to Osteoarthritis: Month 12 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Description: Same event may appear as non-SAE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. The safety analysis set included all participants who received at least one dose of tofacitinib.
Arm/Group | Tofacitinib
All-Cause Mortality (participants affected / at risk) | 2/198
Serious Adverse Events (participants affected / at risk) | 24/198
Other Adverse Events (participants affected / at risk) | 52/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (N=198)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Condition aggravated (General disorders) | 1
Drug ineffective (General disorders) | 7
Pyrexia (General disorders) | 1
Haematotoxicity (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Arthritis bacterial (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Epiglottitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Herpes zoster disseminated (Infections and infestations) | 1
Lower Respiratory Tract infection (Infections and infestations) | 1
Pasteurella infection (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib (N=198)
Uveitis (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Drug ineffective (General disorders) | 13
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Increased Aminotransferases (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bacterial pyelonephritis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 5
Bursitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 9
Cystitis (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Lower Respiratory Tract infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1
Intentional product misuse (Injury, poisoning and procedural complications) | 6
Product dose omission in error (Injury, poisoning and procedural complications) | 1
Product dose omission issue (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hepatic steatosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 1
Haemoglobinuria (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Worsening of already existing skin lesions (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT04079920/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT04079920/SAP_001.pdf